CLINICAL TRIAL: NCT01562678
Title: Liraglutide in Obesity and Diabetes: Identification of CNS Targets Using fMRI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Christos Mantzoros, Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2011P000280
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Results first posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-04

CONDITIONS: Diabetes; Effects of Liraglutide Administration on Brain Activity; Weight Loss; Hunger
Keywords: fMRI; Liraglutide; diabetes; GLP-1
MeSH Terms: conditions — Diabetes Mellitus; Weight Loss | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide (Experimental)
  Interventions: Drug: Liraglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide — In the experimental arm of this randomized, placebo controlled, cross-over, double-blinded study to assess the effects of liraglutide. Subjects will self-inject Liraglutide once per day for 18 days. Subjects will start the treatment with a dose of 0.6 mg for the first week, then 1.2 mg for the second week and 1.8 mg for 3 days in the third week.
  Other Names: victoza
  Arms: Liraglutide
Drug: Placebo — In the placebo arm of this randomized, placebo controlled, cross-over, double-blinded study to assess the effects of liraglutide. Subjects will self-inject placebo once per day for 18 days.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to help us understand the effects of diabetes medication Liraglutide on weight loss and hunger. The investigators have already determined what the highest tolerated dose of Liraglutide is through earlier human research studies. Liraglutide was approved by the FDA in January 2010 for treatment of diabetes.

The investigators will also study the following:

1. The impact of Liraglutide on brain responses to food
2. It's effect on physiological and mental performance
3. If its effect on the brain differs among obese and lean diabetic subjects.

DETAILED DESCRIPTION:
This is a randomized, placebo controlled, cross-over, double-blinded study to assess the effects of liraglutide on brain activation in areas involved in cognitive control and reward during food visualization.

Study participation will span approximately 1.5-2 months. Subjects will learn to self-administer the medication and will have a total of 8 study visits plus one screening visit. The visits will include the following tests/procedures:

1. Vital signs (blood pressure, temperature, heart rate, breathing rate)
2. Height, weight and other body measurements like waist
3. Blood tests
4. Urine pregnancy test (women only)
5. Electrocardiogram (EKG)
6. Medical history
7. Physical exam
8. Body Composition tests
9. Study logs to record food intake and blood sugar
10. functional MRI

We plan to recruit a total of 24 subjects to be treated with placebo and liraglutide. We propose to enroll 12 obese diabetic (type 2) and 12 lean diabetic (type 2) subjects. Equal numbers of men and women will be enrolled and the randomization will block for gender.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be men and women between the ages of 18 and 65. The following table list inclusion criteria for each group (lean diabetic and obese diabetic). Subjects must meet either HbA1c or fasting plasma glucose (FPG) criteria.

Lean diabetic:

BMI: 18-25 kg/m2 HbA1c: < 8.9% Fasting plasma glucose: <250 mg/dL Other inclusion criteria: On dietary modification and/or metformin

Obese diabetic:

BMI: >27 kg/m2 HbA1c: < 8.9% Fasting plasma glucose: <250 mg/dL Other inclusion criteria: On dietary modification and/or metformin

Additionally, women participants must use double barrier methods to prevent pregnancy (diaphragm with intravaginal spermicide, cervical cap, male or female condom with spermicide). If a woman suspects that she has become pregnant at any time or does not use one of the contraceptive methods recommended by the investigator, she must notify the study staff. If a woman becomes pregnant, she will be withdrawn from the study. The study staff will follow the progress of her pregnancy and the birth of her child.

Exclusion Criteria:

1. Uncontrolled diabetes (HbA1c>8.9%, or FPG>250 mg/dL)
2. Women who are breastfeeding, pregnant, or wanting to become pregnant.
3. Women using IUD
4. Any change in the dosage of hormonal contraceptive medications (birth control pills, implanon). Subjects should remain on same medication/ same dose during the time of the entire study.
5. Moderate (creatinine clearance of 30-59 ml/min) and severe renal impairment (creatinine clearance below 30 ml/min) and end-stage renal disease
6. Moderate, or severe hepatic impairment
7. Hypersensitivity to the active substance or any of the excipients in liraglutide
8. History of diabetic ketoacidosis
9. Congestive heart failure
10. Inflammatory conditions like inflammatory bowel disease, Rheumatoid arthritis etc
11. Gastroparesis
12. Pancreatitis
13. Gallstones- as they may cause increased risk of pancreatitis
14. Alcohol consumption- the maximum quantity for men is 140g-210g per week. For women, the range is 84g-140g per week or drinking as consuming no more than two drinks a day for men and one for women. Alcohol can cause increased risk of pancreatitis and hypoglycemia.
15. Untreated thyroid disease like hypothyroidism or hyperthyroidism
16. Subjects taking the following medications: warfarin, steroids (inhaled or systemic due to reduced hypoglycemic effect), and subjects on other hormones (LHRH analogs etc).
17. Subjects on any oral anti-diabetic agent except metformin
18. Personal or family history of MEN II or medullary thyroid cancer
19. Subjects with any type of bioimplant activated by mechanical, electronic, or magnetic means (e.g. cochlear implants, pacemakers, neuron or biostimulators, electronic infusion pumps, etc.)
20. Subjects with any type of metallic implant that could potentially be displaced or damaged during MRI, such as aneurysm clips, metallic skull plates, surgical implants etc. or metal containing tattoos
21. Anxiety and/or claustrophobia
22. Uncontrolled cardiac impairment, circulatory impairment, or inability to perspire (poor thermoregulatory function)
23. Significant sensory or motor impairment
24. Epilepsy, particularly photo-sensitive epilepsy, which may place the individual at a higher risk for adverse events during fMRI scanning with visual stimulation
25. Subjects with neurological problems which may interfere with or complicate testing (e.g. presence of titubation)
26. Body weight above the limitation of the MRI scanning table (330lbs/150 Kg) or body dimensions that could difficult the performance of the scan.
27. Subjects who cannot adhere to the experimental protocol for any reason
28. Anemia with Hgb less than 10
29. Uncontrolled infectious diseases (e.g. HIV, hepatitis, chronic infections etc)
30. Any uncontrolled endocrine condition, e.g Cushing's, Acromegaly, etc
31. Any cancers or lymphoma
32. Eating disorders like anorexia, bulimia
33. Severe hypertriglyceridemia (triglycerides >500 mg/dl)
34. Weight loss surgery or gastrectomy
35. Any changes in medications that affect brain function, e.g. anti-depressants, anti-psychotics, anti-anxiety, anti-seizure medications, antihypertensives etc (subjects should remain on same medication/ same dose during the time of the entire study).
36. Irregular periods, defined as cycle length less than 22 days or more than 40 days.
37. Any change in smoking status.
38. Vegetarians- as food images presented will include numerous non-vegetarian items and thus will not be appealing as high calorie food items.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christos Mantzoros, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Angelidi AM, Kokkinos A, Sanoudou D, Connelly MA, Alexandrou A, Mingrone G, Mantzoros CS. Early metabolomic, lipid and lipoprotein changes in response to medical and surgical therapeutic approaches to obesity. Metabolism. 2023 Jan;138:155346. doi: 10.1016/j.metabol.2022.155346. Epub 2022 Nov 12. PMID 36375643
- [Derived] Farr OM, Sofopoulos M, Tsoukas MA, Dincer F, Thakkar B, Sahin-Efe A, Filippaios A, Bowers J, Srnka A, Gavrieli A, Ko BJ, Liakou C, Kanyuch N, Tseleni-Balafouta S, Mantzoros CS. GLP-1 receptors exist in the parietal cortex, hypothalamus and medulla of human brains and the GLP-1 analogue liraglutide alters brain activity related to highly desirable food cues in individuals with diabetes: a crossover, randomised, placebo-controlled trial. Diabetologia. 2016 May;59(5):954-65. doi: 10.1007/s00125-016-3874-y. Epub 2016 Feb 1. PMID 26831302
- See also: Mantzoros Lab Website — http://www.bidmc.org/Research/Departments/Medicine/Divisions/Endocrinology/Laboratories/MantzorosLab.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Liraglutide First, Then Placebo: 14 participants were randomized to receive Liraglutide and then were cross-overed to receive placebo
- Placebo First, Then Liraglutide: 14 participants were randomized to receive Placebo and then were cross-overed to receive Liraglutide
Period: Overall Study
Arm/Group | Liraglutide First, Then Placebo | Placebo First, Then Liraglutide
Started | 14 | 14
Completed | 8 | 12
Not Completed | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide First, Then Placebo | Placebo First, Then Liraglutide | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (10.5) | 52.5 (10.5) | 52.5 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 7 | 9 | 16
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change Between Highly Desirable vs. Less Desirable Food Cues in the Effect Size of Cortical Activation During Food Visualization
Description: Effect size (region of interest z-scores, derived from z-maps of the brain) shown below is the difference in parietal cortex activation to highly desirable (high fat or high calorie, e.g. cakes, pies, fries) versus less desirable (low fat or low calorie, e.g. vegetables, fruits) food cues for each treatment condition (liraglutide or placebo) at the end of the treatment period.
Time Frame: 18 days of Liraglutide or placebo treatment
Population: Participants with incomplete MRI scans were excluded from the analysis.
Measure: Mean (Standard Error); unit: z-scores of activation in cortex
Groups:
- Liraglutide: Liraglutide: In the experimental phase of this randomized, placebo-controlled, cross-over, double-blinded study to assess the effects of liraglutide, subjects started the treatment with a dose of 0.6 mg for the first week, then 1.2 mg for the second week and 1.8 mg for 3 days in the third week. This sequence may have occurred for their first phase or second phase (placebo was the other phase).
- Placebo: Placebo: In the placebo phase of this randomized, placebo controlled, cross-over, double-blinded study to assess the effects of liraglutide, subjects will self-inject placebo once per day for 18 days. Participants had this first or second (liraglutide was the other phase).
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 18 | 18
z-scores of activation in cortex | -0.42 (0.27) | 0.53 (0.37)

ADVERSE EVENTS:
Time Frame: Throughout the study (4 visits in each phase of liraglutide and placebo).
Description: There was a systematic assessment of adverse events at each visit (Days 0, 7, 14, and 17) by an MD who asked detailed medical questions and did a physical exam, plus through the use of visual analog scales administered 3 times per day where participants answered on a 10cm line questions such as "How nauseous do you feel right now?"
Groups:
- Liraglutide: 14 participants were randomized to receive Liraglutide and then were cross-overed to receive placebo and 14 participants were randomized to receive Placebo and then were cross-overed to receive Liraglutide
- Placebo: 14 participants were randomized to receive Placebo and then were cross-overed to receive Liraglutide and 14 participants were randomized to receive Liraglutide and then were cross-overed to receive placebo
Arm/Group | Liraglutide | Placebo
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 7/28 | 7/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=28) | Placebo (N=28)
Nausea (Gastrointestinal disorders) | 7 (7) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No